CLINICAL TRIAL: NCT02543281
Title: Adaptive CRT Effect on Electrical Dyssynchrony
Acronym: aCRT-ELSYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larisa Tereshchenko (Other)
Responsible Party: Sponsor-Investigator, Larisa Tereshchenko, Assistant Professor, Department of Medicine, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-11299
Record Dates: First submitted 2015-09-01; First posted 2015-09-07 (Estimated); Results first posted 2023-11-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cardiomyopathy; Heart Failure; Left Bundle Branch Block
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aCRT Off (Active Comparator): The adaptive CRT algorithm will be turned off for the CRT device implanted in the patients in this arm.
  Interventions: Device: Conventional Cardiac Resynchronization Therapy
- aCRT On (Experimental): The adaptive CRT algorithm will be turned on for the CRT device implanted in the patients in this arm.
  Interventions: Device: Adaptive cardiac resynchronization therapy
- Registry arm (No Intervention): Participants who are not eligible for the randomization because of the implantation of the device that is not capable of delivering aCRT. The team of clinical care providers makes such a clinical decision acting in the patient's best interests.

INTERVENTIONS:
Device: Adaptive cardiac resynchronization therapy — The adaptive cardiac resynchronization therapy (aCRT) algorithm works by sometimes giving stimulation to only the left side of the heart, rather than to both sides, depending on how it senses the heart is functioning.
  Other Names: aCRT
  Arms: aCRT On
Device: Conventional Cardiac Resynchronization Therapy — CRT without the adaptive algorithm works by giving stimulation to both sides of the heart.
  Other Names: CRT
  Arms: aCRT Off

SUMMARY:
The purpose of this study is to better understand how adaptive cardiac resynchronization therapy (aCRT) might benefit patients. aCRT works by sometimes giving stimulation to only the left side of the heart, rather than to both sides, depending on how it senses the heart is functioning. CRT without the adaptive algorithm works by giving stimulation to both sides of the heart. aCRT has already been approved by the FDA and is being used in patients now, but it is not clear which patients it should be used in compared to normal CRT. This study will include patients who are already scheduled to get a CRT device. The investigators will then randomize patients to the aCRT study arm or to the CRT study arm. After 6 months, the investigators will assess the electrical activity of the patients' hearts. After this time, the patient and their doctors will be able to decide if they would like to change the type CRT they have been designated.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a standard class I or class II indications for CRT-P or CRT-D implantation in accordance with ACC/AHA/HRS guidelines (2012 ACCF/AHA/HRS Focused Update Incorporated Into the ACCF/AHA/HRS 2008 Guidelines for Device-Based Therapy of Cardiac Rhythm Abnormalities)2.At least 18 years of age at the time of consent
* Is willing and able to comply with the protocol

Exclusion Criteria:

* Chronic atrial arrhythmias defined as: "Atrial fibrillation is permanent when it has resisted all attempts to restore sinus rhythm or when the physician and patient decide that no such attempt should be made."
* Patient has ever had a previous or has an existing CRT system, ICD, or pacemaker.
* GFR <30ml/min
* Patient has had unstable angina, acute myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty within 30 days prior to study enrollment
* Patient has primary valvular disease and is indicated for valve repair or replacement
* Patient is enrolled in ≥1 concurrent studies that would confound the study results (any other interventional trial)
* Patient is pregnant or of childbearing potential and not on a reliable form of birth control. All women of child-bearing potential must undergo a pregnancy test.
* Patient status post heart transplant
* Patient has been classified as NYHA functional class IV within 3 months prior to study enrollment
* concomitant conditions other than cardiac diseases that were associated with a higher likelihood of death during 1 year after enrollment
* Patient, legal guardian or authorized representative is unable or unwilling to cooperate or give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Tereshchenko, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Haq KT, Rogovoy NM, Thomas JA, Hamilton C, Lutz KJ, Wirth A, Bender AB, German DM, Przybylowicz R, van Dam P, Dewland TA, Dalouk K, Stecker E, Nazer B, Jessel PM, MacMurdy KS, Zarraga IGE, Beitinjaneh B, Henrikson CA, Raitt M, Fuss C, Ferencik M, Tereshchenko LG. Adaptive Cardiac Resynchronization Therapy Effect on Electrical Dyssynchrony (aCRT-ELSYNC): A randomized controlled trial. Heart Rhythm O2. 2021 Jun 29;2(4):374-381. doi: 10.1016/j.hroo.2021.06.006. eCollection 2021 Aug. PMID 34430943

RESULTS

PARTICIPANT FLOW:
Groups:
- Registry: Participants who were not eligible for the randomization because of the implantation of the device that was not capable of delivering aCRT. The team of clinical care providers made such a clinical decision acting in the best interests of a patient.
Period: Overall Study
Arm/Group | aCRT Off | aCRT On | Registry
Started | 15 | 12 | 5
Completed | 15 | 12 | 4
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- aCRT Off: The adaptive CRT algorithm turned off for the CRT device implanted in the patients in this arm.
  Conventional Cardiac Resynchronization Therapy: CRT without the adaptive algorithm works by giving stimulation to both sides of the heart.
- aCRT On: The adaptive CRT algorithm turned on for the CRT device implanted in the patients in this arm.
  Adaptive cardiac resynchronization therapy: The adaptive cardiac resynchronization therapy (aCRT) algorithm works by sometimes giving stimulation to only the left side of the heart, rather than to both sides, depending on how it senses the heart is functioning.
- Total: Total of all reporting groups
Arm/Group | aCRT Off | aCRT On | Registry | Total
Number analyzed (Participants) | 15 | 12 | 5 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (12.2) | 62.2 (10.3) | 67.3 (13.6) | 64.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 11
  Male | 10 | 8 | 3 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Non-Hispanic White | 15 | 11 | 5 | 31
  Race and Ethnicity: Non-White or Hispanic | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 5 | 32
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Percentage of Left Ventricular EF] — Percentage of Left Ventricular Ejection Fraction
  Percentage of Left Ventricular EF | 26 (8.6) | 29.7 (7.5) | 32.3 (6.4) | 28.4 (8.0)
Ischemic cardiomyopathy [Count of Participants; unit: Participants]
  Ischemic cardiomyopathy | 9 | 5 | 3 | 17
  Non-ischemic cardiomyopathy | 6 | 7 | 2 | 15
QRS duration [Mean (Standard Deviation); unit: ms] | 151.3 (24.3) | 160.6 (19.0) | 153.1 (20.9) | 155.1 (20.9)
Left Bundle Branch Block [Count of Participants; unit: Participants]
  Left Bundle Branch Block (strict criteria) | 1 | 4 | 0 | 5
  Non - Left Bundle Branch Block | 14 | 8 | 5 | 27
NYHA Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification graded patients based on their symptoms and limitations of physical activity. Overall, there are four classes. The higher class the worse.
  Class III is worse than Class II. Class II patients experience slight limitations in physical activity. Ordinary physical activity results in fatigue, palpitation, and shortness of breath.
  Class III patients experience marked limitations in physical activity. Less than ordinary physical activity activity causes fatigue, palpitation, and shortness of breath.
  Participants
    NYHA Class II (less severe) | 9 | 8 | 4 | 21
    NYHA Class III (more severe) | 6 | 4 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Ventricular Electrical Uncoupling (VEU), Calculated as the Difference in Difference Between the Mean Left Ventricular (LV) and Right Ventricular (RV) Activation Times.
Description: LV and RV activation time values were measured on reconstructed epicardial activation maps at baseline and 6 months post-CRT. Positive VEU indicated LV uncoupling (delay) from the RV, whereas negative VEU indicated RV uncoupling (delay) from the LV. Difference in difference (change in VEU from baseline to 6 months post-CRT) is reported as the primary outcome.
Time Frame: baseline and 6 months after device implantation
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | aCRT Off | aCRT On | Registry
Number analyzed (Participants) | 15 | 12 | 4
ms | 21.4 [-30.0 to 49.9] | 18.9 [4.3 to 29.2] | 6.0 [-8.0 to 11.6]

2. Secondary Outcome: Change in 6-minute Walk Distance 6 Months Post CRT
Description: Change in 6-minute walk distance 6 months post CRT as compared to baseline
Time Frame: baseline and 6 months after device implantation
Measure: Median (Inter-Quartile Range); unit: m
Arm/Group | aCRT Off | aCRT On | Registry
Number analyzed (Participants) | 15 | 12 | 4
m | 18 [-12 to 41] | -19 [-76 to 57] | 141 [66 to 215]

3. Secondary Outcome: Change in MLHFQ Total Score
Description: Change in Minnesota Living with Heart Failure Questionnaire (MLHFQ) total score 6 months post-CRT as compared to baseline. The total MLHFQ score range from 0 (zero; the best health) to 105 (the worst health). Higher MLHFQ values represent worse health. Negative values of the change in total MLHFQ score mean the total MLHFQ score decreased six months after device implantation compared to baseline (improvement).
Time Frame: baseline and 6 months after device implantation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | aCRT Off | aCRT On | Registry
Number analyzed (Participants) | 15 | 12 | 4
units on a scale | -20 [-30 to -4] | -7 [-15 to 0.5] | -28 [-43 to -9]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | aCRT Off | aCRT On | Registry
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT02543281/Prot_SAP_000.pdf